CLINICAL TRIAL: NCT03741400
Title: Virtual Reality Glove for Hand and Arm Rehabilitation After Stroke
Acronym: vREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: NEOFECT Rehabilitation Solutions (Other)
Responsible Party: Principal Investigator, Maarten Lansberg, Associate Professor, Neurology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46423
Record Dates: First submitted 2018-10-17; First posted 2018-11-14 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Acute; Cerebral Infarction
Keywords: motor weakness; rehabilitation
MeSH Terms: conditions — Stroke; Cerebral Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor that will be performing the interval assessments will be blinded to treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Occupational Therapy + Smart Glove (Experimental): Subjects randomized to this arm will be expected to use the Neofect Rapael Smart Glove for a minimum of 20-30 minutes per day, 5 days per week, in addition to prescribed occupational therapy.
  Interventions: Device: Neofect RAPAEL Smart Glove
- Standard Occupational Therapy (No Intervention): Subjects in the control arm will undergo standard of care occupational therapy as prescribed by their care team.

INTERVENTIONS:
Device: Neofect RAPAEL Smart Glove — The Neofect Rapael Smart Glove is a biofeedback system designed for upper extremity rehabilitation in stroke survivors. It includes a glove-shaped sensor device and a software application.
  Arms: Standard Occupational Therapy + Smart Glove

SUMMARY:
The Virtual Reality Glove for Hand and Arm Rehabilitation (vREHAB) trial is a randomized, controlled, phase 3 trial aiming to evaluate the safety, usability, and efficacy of a virtual reality biofeedback system (Neofect RAPAEL Smart Glove) to promote recovery of distal arm and hand function in the acute and subacute period after stroke, as compared to standard of care therapy. The aims of the study is to demonstrate:

1. the effect of Smart Glove use on functional recovery, in addition to standard of care rehabilitation therapy.
2. the feasibility of increasing the dose of rehabilitation in acute stroke patients with the Smart Glove.
3. the effect of Smart Glove use on quality of life.

DETAILED DESCRIPTION:
The Neofect Smart Glove is a commercially available, non-invasive biofeedback based system for distal upper extremity rehabilitation. The Smart Glove is very lightweight and allows for easy movement of all distal upper extremity joints. It consists of a glove-shaped sensor device and a software application which can be used with either a large screen or a portable tablet. The system includes multiple Activities of Daily Living (ADL)-based training games, and the system tracks the motion and posture of the wearer's distal limb as they participate. Games can be selected to focus on certain movements (such as forearm pronation/supination, wrist flexion/extension, finger flexion/extension, etc.) based on the needs of the wearer. The software includes a smart learning algorithm, in which the computer automatically adjusts to the optimal level of difficulty to balance challenge and motivation. After initial set-up, the device requires no therapist supervision to use.

Patients will be eligible for the study if they have had an ischemic or hemorrhagic stroke and (2) have impaired arm/hand function secondary to the stroke (see below for specific inclusion and exclusion criteria). We will recruit eligible patients from acute care hospitals, acute rehabilitation units, and outpatient facilities. Enrolled patients will be randomized (1:1 ratio) to standard rehabilitation therapy versus standard rehabilitation therapy plus Smart Glove use. All patients will be allowed to participate in any scheduled outpatient rehabilitation during the study.

The study consists of a 12-week intervention period and a 12-week follow-up period. During the 12-week intervention period all patients will receive their usual rehabilitation therapy, with their therapists documenting rehabilitation dose in a journal provided at the start of the study. In addition, subjects randomized to the Smart Glove therapy arm will be provided with a Smart Glove system, which includes the glove and tablet. Subjects will be instructed to use the system for at least one session per day for 5 days per week during the 12-week intervention period. Participants will present for in-person visits on weeks 6, 12, and 24 for blinded assessments by study coordinators. At the completion of the intervention period, subjects will return the Smart Glove and subjects in both arms of the study will only receive usual care during the 12-week follow-up period. Subjects will have a final assessment at week 24 (12 weeks after completing the intervention) to assess for persistence of effect.

All efficacy analyses are analyzed under the intention to treat principle. The primary efficacy outcome is the change in score on the Jebsen Taylor Hand Test between baseline and week 12. Secondary efficacy endpoints are changes in scores on the upper extremity Fugl-Meyer Scale, Stroke Impact Scale, and total dose of rehabilitation received during the 24-week intervention period. Persistence of the treatment effect will be tested by comparing changes in scores on the Jebsen Taylor Hand Test and Fugl-Meyer upper extremity score at 24 weeks between treatment groups

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of ischemic or hemorrhagic stroke prior to enrollment.
* unilateral hand/arm weakness from stroke with indication for upper limb rehabilitation therapy.
* ability to successfully play 2 out 4 pre-selected test games with the Smart Glove. The test specific games and criteria for passing are as follows:

  * Pour the wine (Pronation/Supination): make 5 pours in first 1 minute
  * Snow Ball Fight (Wrist Flexion/Extension w/ gravity eliminated): take down 3 objects in first 1 minute
  * Scrub the Floor (Wrist Radial/Ulnar deviation w/ gravity eliminated): scrub the floor 5 times in first 1 minute
  * Float the Fish (Finger Flexion/Extension): make 50 meters with 3 or less bumps in first 3 minutes

Exclusion Criteria:

* Age <18 years
* history of visually provoked seizures
* psychological disorder that could impede participation
* pre-existing neurologic disorder which causes significant deficits in arm/hand function (e.g. Parkinson's disease, peripheral neuropathy, etc.)
* severe receptive aphasia which results in inability to participate with the Smart Glove.
* cognitive impairment which results in inability to participate with the Smart Glove.
* severe pain impeding upper extremity rehabilitation and use of the Smart Glove
* limited life-expectancy which makes it unlikely that patient will be able to complete the 24-week follow-up visit
* any medical or other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten G Lansberg, MD, Principal Investigator — Stanford University
Locations (4):
- United States (3):
  - Stanford University, Palo Alto, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Intermountain Healthcare, Salt Lake City, Utah
- UZ Leuven, Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Occupational Therapy: Participants in the control arm undergo standard of care occupational therapy as prescribed by their care team.
- Standard Occupational Therapy + Smart Glove: Participants randomized to this arm use the Neofect Rapael Smart Glove for a minimum of 20-30 minutes per day, 5 days per week, in addition to prescribed occupational therapy.
Period: Overall Study
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
Started | 30 | 30
Completed | 24 | 18
Not Completed | 6 | 12

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [55 to 72] | 59 [45 to 65] | 60 [50 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 17 | 11 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 21 | 14 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 3 | 9
  Black or African American | 0 | 1 | 1
  White | 16 | 11 | 27
  Other | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 12 | 28
  Belgium | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Impairment, Jebsen Taylor Hand Function Test
Description: The change in scores on the Jebsen-Taylor hand function test (JTHFT) from baseline to twelve weeks (in seconds) was compared between treatment groups.
  The JTHFT is a standardized and objective measure of hand functions commonly used in activities of daily living (ADLs). The test consists of seven subtests separated into fine (JTHFT-Fine) and gross (JTHFT-Gross) motor tasks. Fine motor tasks include writing, simulated page turning, lifting small objects, and simulated feeding. Gross motor tasks include stacking checkers, lifting large light objects, and lifting large heavy objects. The score was calculated as the total number of seconds to perform the tasks, with a lower score indicating better function. Patients who could not complete a task within 90 seconds were assigned a maximum score of 90 seconds for that task. Therefore, the maximum score was 360 sec for the JTHFT-Fine, 270 sec for the JTHFT-Gross, and 630 sec for the JTHFT-Total.
Time Frame: baseline, 12 weeks
Population: Participants who completed the protocol.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
Number analyzed (Participants) | 24 | 18
seconds
  Baseline-Total | 119 [92 to 176] | 181 [150 to 286]
  Change at week 12-Total | -69 [-129 to -20] | -64 [-151 to -26]
  Baseline-Fine | 87 [65 to 126] | 131 [97 to 185]
  Change at week 12-Fine | -37 [-99 to -8] | -35 [-93 to -16]
  Baseline-Gross | 30 [23 to 44] | 59 [50 to 84]
  Change at week 12-Gross | -23 [-92 to -5] | -31 [-49 to -8]
Statistical Analysis 1: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis of change in total seconds; Test type: Other; p = 0.88, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS
Statistical Analysis 2: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis of change in fine motor skill assessment; Test type: Other; p = 0.99, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS
Statistical Analysis 3: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis of change in gross motor skills assessment; Test type: Other; p = 0.80, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS

2. Secondary Outcome: Change in Functional Impairment, Upper Extremity Fugl-Meyer Assessment
Description: The change in scores on the Upper Extremity Fugl-Meyer [0-66, with higher score meaning better motor function] test from baseline to twelve weeks will be compared between treatment groups. The test measures reflex activity, selective movement, and coordination of the hand, wrist, forearm, elbow, and shoulder.
Time Frame: baseline, 12 weeks
Population: Participants who completed the protocol
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
Number analyzed (Participants) | 24 | 18
score on a scale
  Baseline | 55 [51 to 57] | 46 [40 to 54]
  Change at week 12 | 8 [2 to 13] | 8 [5 to 17]
Statistical Analysis 1: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Test type: Other; p = 0.61, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS

3. Secondary Outcome: Persistence of Treatment Effects at 24 Weeks in Jebsen Taylor Hand Function Test
Description: The change in scores on the Jebsen-Taylor hand function test from baseline to twenty-four weeks (in seconds) was compared between treatment groups.
  The JTHFT is a standardized and objective measure of hand functions commonly used in activities of daily living (ADLs). The test consists of seven subtests separated into fine (JTHFT-Fine) and gross (JTHFT-Gross) motor tasks. Fine motor tasks include writing, simulated page turning, lifting small objects, and simulated feeding. Gross motor tasks include stacking checkers, lifting large light objects, and lifting large heavy objects. The score was calculated as the total number of seconds to perform the tasks, with a lower score indicating better function. Patients who could not complete a task within 90 seconds were assigned a maximum score of 90 seconds for that task. Therefore, the maximum score was 360 sec for the JTHFT-Fine, 270 sec for the JTHFT-Gross, and 630 sec for the JTHFT-Total.
Time Frame: baseline, 24 weeks
Population: Participants who completed the protocol.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
Number analyzed (Participants) | 24 | 18
seconds
  Baseline-Total | 119 [92 to 176] | 181 [150 to 286]
  Change at week 24-Total | -47 [-107 to -17] | -82 [-145 to -45]
  Baseline-Fine | 87 [65 to 126] | 131 [97 to 185]
  Change at week 24-Fine | -37 [-99 to -8] | -35 [-93 to -16]
  Baseline-Gross Baseline-Gross | 30 [23 to 44] | 59 [50 to 84]
  Change at week 24-Gross | -16 [-38 to -3] | -33 [-58 to -23]
Statistical Analysis 1: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis of change in total seconds; Test type: Other; p = 0.47, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS
Statistical Analysis 2: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis of change in fine motor skill assessment; Test type: Other; p = 0.55, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS
Statistical Analysis 3: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis of change in gross motor skills assessment; Test type: Other; p = 0.38, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS

4. Secondary Outcome: Persistence of Treatment Effects at 24 Weeks in Upper Extremity Fugl-Meyer Test
Description: Change in scores in Upper Extremity Fugl-Meyer [0-66, with higher score meaning better motor function] test between baseline and 24 weeks will be compared between treatment groups. The test measures reflex activity, selective movement, and coordination of the hand, wrist, forearm, elbow, and shoulder.
Time Frame: baseline, 24 weeks
Population: Participants who completed the protocol
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
Number analyzed (Participants) | 24 | 18
score on a scale
  Baseline | 55 [51 to 57] | 46 [40 to 54]
  Change at week 24 | 7 [0 to 13] | 11 [6 to 19]
Statistical Analysis 1: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Test type: Other; p = 0.24, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS

5. Secondary Outcome: Total Dose of Upper Extremity Rehabilitation
Description: Total dose (minutes) of all upper extremity rehabilitation therapy, including Smart Glove therapy, received during the 12-week intervention period will be compared between treatment groups.
Time Frame: 12 weeks
Population: Participants who completed the protocol and with available data.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
Number analyzed (Participants) | 22 | 18
minutes | 584 [300 to 1375] | 1434 [464 to 2520]
Statistical Analysis 1: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Test type: Other; p = 0.18, Mann-Whitney U test — A priori threshold for statistical significance, 0.05

6. Secondary Outcome: Self-rated Stroke-related Disability Between Each Treatment Group
Description: Domain scores (0-100, with 100 being better self-rated function in each of: strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion, memory/thinking, and participation) on the Stroke Impact Scale will be compared between treatment groups at 12 weeks and at 24 weeks.
Time Frame: Weeks 12 and 24
Population: Participants with available data at the respective time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
Number analyzed (Participants) | 24 | 17
score on a scale
  Week 12 | 63 [38 to 88] | 65 [40 to 85]
  Week 24 | 75 [60 to 100] | 82.5 [60 to 85]
Statistical Analysis 1: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis at week 12; Test type: Other; p = 0.926, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS
Statistical Analysis 2: Comparison: Standard Occupational Therapy vs Standard Occupational Therapy + Smart Glove; Analysis at week 24; Test type: Other; p = 0.828, ANCOVA — A priori threshold for statistical significance, 0.05; Nonparametric ANCOVA using Quade's test with adjustments for age, sex, and NIHSS

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Standard Occupational Therapy | Standard Occupational Therapy + Smart Glove
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 7/30 | 9/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Occupational Therapy (N=30) | Standard Occupational Therapy + Smart Glove (N=30)
Stroke (Vascular disorders) | 0 | 1 — Not related to study treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Occupational Therapy (N=30) | Standard Occupational Therapy + Smart Glove (N=30)
atrial fibrilation (Cardiac disorders) | 0 | 2 — Not related to study treatment
compression fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 — Not related to study treatment
COVID-19 (Infections and infestations) | 0 | 1 — Not related to study treatment
cystitis (Infections and infestations) | 1 | 0 — Not related to study treatment
dehydration (General disorders) | 0 | 1 — Not related to study treatment
diarrhea (Gastrointestinal disorders) | 1 | 0 — Not related to study treatment
dizziness (Nervous system disorders) | 1 | 0 — Not related to study treatment
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not related to study treatment
ennui (General disorders) | 0 | 1 — Not related to study treatment
eyelid injury (Eye disorders) | 1 | 0 — Not related to study treatment
fall (Injury, poisoning and procedural complications) | 1 | 2 — Not related to study treatment
fever (Infections and infestations) | 1 | 0 — Not related to study treatment
headache (Nervous system disorders) | 1 | 1 — Not related to study treatment
hypertension (Cardiac disorders) | 0 | 1 — Not related to study treatment
hypokalemia (Metabolism and nutrition disorders) | 0 | 1 — Not related to study treatment
hypotension (Cardiac disorders) | 1 | 1 — Not related to study treatment
inversion trauma ankle (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to study treatment
loss of balance (Nervous system disorders) | 0 | 1 — Not related to study treatment
multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Not related to study treatment
pain (General disorders) | 1 | 2 — Not related to study treatment
phalanx fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 — Not related to study treatment
pneumonia (Infections and infestations) | 0 | 1 — Not related to study treatment
reduced strength (Musculoskeletal and connective tissue disorders) | 0 | 1 — Not related to study treatment
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Not related to study treatment
syncope (Cardiac disorders) | 0 | 1 — Not related to study treatment
upper extremity stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 — Not related to study treatment
urinary retention (Renal and urinary disorders) | 0 | 1 — Not related to study treatment
urinary tract infection (Renal and urinary disorders) | 0 | 1 — Not related to study treatment
weight loss (General disorders) | 1 | 0 — Not related to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03741400/Prot_SAP_000.pdf